CLINICAL TRIAL: NCT03585504
Title: A Randomized Controlled Trial of Immediate Versus Delayed Insertion of Implanon in Postpartum Adolescents
Brief Title: Immediate Versus Delayed Insertion of Implanon in Postpartum Adolescents
Acronym: Implanon
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: American College of Obstetricians and Gynecologists (Other); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HR #19133
Record Dates: First submitted 2018-05-10; First posted 2018-07-13 (Actual); Results first posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Contraceptive Usage
Keywords: Implanon; Bleeding Acceptability; Contraceptive Implant; Adolescent Pregnancy Prevention; Post Partum Insertion of Implanon
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: participants were randomized to receive a contraceptive implant before hospital discharge or at their six week postpartum visit
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients will undergo etonogestrel contraceptive implant insertion prior to hospital discharge per package instructions.
  Interventions: Drug: Etonogestrel contraceptive implant
- Control Group (Active Comparator): These patients will receive an appointment to undergo etonogestrel contraceptive implant insertion at the postpartum visit occuring approximately six weeks after delivery as is standard care in our institution.
  Interventions: Drug: Etonogestrel contraceptive implant

INTERVENTIONS:
Drug: Etonogestrel contraceptive implant — Etonogestrel contraceptive implant

SUMMARY:
The specific aim of this study is to evaluate whether insertion of a long-acting contraceptive implant in postpartum adolescents prior to hospital discharge increases use of this highly effective contraception during the first twelve months postpartum among adolescents who elect Implanon® as their preferred method of contraception. Additionally, this study aims to compare the acceptability of bleeding in postpartum adolescents who have an etonogestrel contraceptive implant prior to discharge versus those with insertion at the six week postpartum visit. The investigators will evaluate the acceptability of bleeding rather than collect prospective diaries because the investigators feel subjective perceptions of bleeding impact contraceptive continuation more than quantitative differences in bleeding.

DETAILED DESCRIPTION:
Study Design and Subject Recruitment The investigators propose a prospective randomized trial comparing immediate postpartum insertion of Implanon® versus insertion at the standard six week postpartum visit in adolescents. Recruitment will occur on our postpartum ward.

The study coordinator will approach all eligible women on the postpartum ward to offer comprehensive contraceptive counseling including information about Implanon® as well as other methods. Those who choose Implanon® will be screened for eligibility and consented for participation in the study. If a subject is under 18 years of age, the investigators will obtain parental consent from at least one parent or legal guardian as well as assent from the adolescent participant according to our IRB guidelines. Those who are not interested in participation will be provided with a standard postpartum appointment for insertion. Based on our volume of adolescent deliveries, the investigators anticipate to complete enrollment within 1 year and follow-up within two years.

Inclusion and Exclusion Criteria Women will be eligible for enrollment if they are 21 years old or younger, English or Spanish speaking, less than 120 hours (5 days) postpartum after either vaginal or cesarean delivery, primiparous or multiparous, and breast and/or bottle-feeding. Women will be excluded from enrollment if they have contraindications to Implanon® insertion including current or prior thrombo-embolic disease, liver disease, hypersensitivity to components of Implanon®, or are using medications such as rifampin, phenytoin, or carbamazepine that increase metabolism of steroid hormones. Women will also be excluded if they indicate unwillingness to continue follow-up for one year.

Randomization After consent is obtained, each participant will be randomized to one of two groups. The study coordinator will open opaque sealed envelopes containing group assignment in sequence. The envelopes will be prepared by a research staff member not involved in recruitment or analysis prior to start of enrollment. The randomization scheme will utilize permuted blocks of sizes four and six. The intervention group will undergo Implanon® insertion prior to hospital discharge per package instructions. For those randomized to this group, the study coordinator will notify the physician on call to ensure insertion prior to discharge. This will not prolong hospital stay. The control group will receive an appointment to undergo Implanon® insertion at the postpartum visit occurring approximately six weeks after delivery as is standard care in our institution. In addition to standard counseling to avoid sexual intercourse for six weeks, all participants will be counseled about condom use for prevention of both sexually transmitted infections and pregnancy.

Follow-up At the time of enrollment, each participant will complete a questionnaire to collect information about sociodemographic characteristics, sexual and reproductive history, contraceptive history, bleeding expectations, breast feeding intentions, and prior sexual education experiences. Each participant will be provided with a notice of study participation to give their provider at their postpartum follow-up visit but there will not be contact between study staff and participants at the six week postpartum visit. Each participant will be contacted by telephone at three, six, and twelve months postpartum. Follow-up questionnaires will be administered at this time to assess use of Implanon® since delivery, use of other highly effective and less effective contraceptive methods, the acceptability of bleeding experiences, and the prevalence and duration of breastfeeding.

Outcomes

* Primary Outcome is the proportion of participants in each group using Implanon® at six months.
* Secondary Outcomes Contraceptive Use and Pregnancy
* Proportion of participants using Implanon at three months
* Proportion of participants using Implanon at twelve months
* Proportion of participants using another highly effective method at three, six, and twelve months.

(Intrauterine contraception and sterilization will be considered highly effective in this study.)

* Proportion of participants using a less effective method at three, six, and twelve months. (DMPA, combined hormonal oral contraception, vaginal ring, transdermal patch, progestin only pills, and barrier methods will be considered less effective methods in this study.)
* Proportion of participants practicing abstinence at three, six, and twelve months.
* Proportion of participants using no contraceptive method at three, six, and twelve months.
* Reasons for non-use of Implanon at three, six, and twelve months.
* Reasons for non-use of any method at three, six, and twelve months.
* Pregnancy rate in each group at twelve months.

  o Bleeding Acceptability
* Bleeding expectations prior to insertion of Implanon
* Comparison of bleeding perceptions to pre-insertion expectations
* Proportion of participants who cite bleeding irregularities as a reason for non-use at three, six, and twelve months
* Satisfaction with bleeding on Likert scale

  o Overall Acceptability 5 of 12
* Proportion at three, six, and twelve months willing to use Implanon again after another delivery
* Proportion at three, six, and twelve months willing to recommend Implanon to a friend

  o Breast Feeding
* Proportion of participants in each group planning to breastfeed at time of enrollment
* Proportion of participants breast feeding at three, six, and twelve months
* Duration of breast feeding in weeks by participant report

ELIGIBILITY:
Inclusion Criteria:

* ages 15-21
* women
* english or spanish speaking
* less than 120 hours post partum

Exclusion Criteria:

* women who are breastfeeding
* contraindications to Implanon® insertion including current or prior thrombo-embolic disease, liver disease, hypersensitivity to components of Implanon®, or are using medications such as rifampin, phenytoin, or carbamazepine that increase metabolism of steroid hormones.
* indicate unwillingness to continue follow-up for one year.

Ages: 15 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Dempsey, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Sothornwit J, Kaewrudee S, Lumbiganon P, Pattanittum P, Averbach SH. Immediate versus delayed postpartum insertion of contraceptive implant and IUD for contraception. Cochrane Database Syst Rev. 2022 Oct 27;10(10):CD011913. doi: 10.1002/14651858.CD011913.pub3. PMID 36302159

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 41 | 40
Completed | 15 | 11
Not Completed | 26 | 29
Not completed — Lost to Follow-up | 26 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Continuous [Median (Standard Deviation); unit: years] — Population: Age was not recorded in the baseline questionnaire.
  years
    number analyzed (Participants) | 15 | 11 | 26
    (all) | 18.93 (1.64) | 19.64 (1.03) | 19.24 (1.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 40 | 81
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 30 | 31 | 61
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 41 | 40 | 81

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Contraceptive Implant Continuation at Six Months Postpartum
Description: We compare the number of participants continuing the implant at six months in each group.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 15 | 11
Participants | 15 | 7

2. Secondary Outcome: Number of Participants That Reported They Were Somewhat or Very Satisfied With Their Subjective Bleeding Experience at Six Months Postpartum.
Description: Compare the number of participants who reported that they were somewhat or very satisfied with their subjective bleeding experience at six months postpartum in each group. Each participant was asked, "Please indicate your overall level of satisfaction with your bleeding." The response options were "very satisfied", "somewhat satisfied", "somewhat dissatisfied", and "very dissatisfied". The outcome measure was treated as a categorical variable.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 15 | 11
Participants | 10 | 8

3. Secondary Outcome: Number of Participants Who Reported That They Were Somewhat or Very Satisfied With the Contraceptive Implant at Six Months Postpartum.
Description: Comparison of the number of participants in each group who report that they were somewhat or very satisfied with their contraceptive method choice at six months postpartum in each group. Participants were asked, " How would you rate your overall satisfaction with implanon?" The response options were "very satisfied", "somewhat satisfied", "somewhat dissatisfied", and "very dissatisfied". The outcome measure was treated as a categorical variable.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 15 | 11
Participants | 14 | 6

ADVERSE EVENTS:
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/11
Other Adverse Events (participants affected / at risk) | 0/15 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No